CLINICAL TRIAL: NCT00807794
Title: Phase I Evaluation of the Pharmacokinetics, Pharmacodynamics and Safety of Different Doses of MEDI-507 in the Prevention of Acute Renal Allograft Rejection
Brief Title: A Safety Clinical Trial of Different Doses of MEDI-507 in the Prevention of Acute Renal Allograft Rejection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: J. Bruce McClain, M.D., Medimmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP027
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — siplizumab

ARMS (5):
- 1 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 2 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 3 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 4 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507
- 5 (Experimental): MEDI-507
  Interventions: Drug: MEDI-507

INTERVENTIONS:
Drug: MEDI-507 — 0.012 mg/kg dose given twice between 60 to 72 hours apart
  Arms: 1
Drug: MEDI-507 — 0.06 mg/kg dose given twice between 60 to 72 hours apart
  Arms: 2
Drug: MEDI-507 — 0.12 mg/kg dose given twice between 60 to 72 hours apart
  Arms: 3
Drug: MEDI-507 — 0.24 mg/kg dose given twice between 60 to 72 hours apart (supplemental)
  Arms: 4
Drug: MEDI-507 — 0.50 mg/kg dose given twice between 60 to 72 hours apart (supplemental)
  Arms: 5

SUMMARY:
To evaluate the clinical safety of different doses of MEDI-507 through day 33.

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic characteristics of MEDI-507 given in dose intervals.

ELIGIBILITY:
Inclusion Criteria:

* Renal allograft recipients receiving their first or second allograft
* Age over 18
* Maintained on conventional immunosuppression
* Completed informed consent document

Exclusion Criteria:

* Known hypersensitivity to MEDI-507
* More than two renal allografts
* Moribund and unlikely (in the opinion of the investigator) to survive the duration of the trial
* Simultaneous use of other investigational agents (this does not include the use of licensed agents for indications not listed in the package insert)
* Any of the following clinical settings or diagnoses posttransplant:

pregnancy or nursing mother: Ø Human Immunodeficiency Virus infection Ø hemodialysis or chronic peritoneal dialysis Ø use of a ventilator Ø hyperacute rejection

* Having received OKT3, tacrolimus, or antilymphocyte globulin during the current allograft
* Less than 10 ml/hr average urine output over 4 hours since the end of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1997-02; Primary Completion 1997-11 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical safety of MEDI-507. Each adverse event will be reported by severity grade, relationship to study drug, organ system, and need for medical intervention. | Day 33

SECONDARY OUTCOMES:
To collect initial pharmacokinetic parameters, the incidence and time to first episode of acute rejection, the number of episodes of rejection and graft survival. | Day 33

CONTACTS AND LOCATIONS:
Overall Officials: J. Bruce McClain, M.D., Study Director — MedImmune LLC
Locations (4):
- United States (4):
  - Yale University School of Medicine, New Haven, Connecticut
  - Indiana University, Bloomington, Indiana
  - San Antonio Community Hospital, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia